CLINICAL TRIAL: NCT00424060
Title: Phase II Study of ZK 219477 in Patients With Recurrent Glioblastoma
Brief Title: Epothilone ZK-219477 in Treating Patients With Recurrent Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-26061; EORTC-26061; EUDRACT-2006-001659-37; SPRI-EORTC-26061
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; recurrent adult brain tumor; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Brain Neoplasms; Gliosarcoma | interventions — sagopilone; In Situ Hybridization, Fluorescence; Gene Expression Profiling; Immunohistochemistry

INTERVENTIONS:
Drug: sagopilone
Genetic: fluorescence in situ hybridization
Genetic: gene expression analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as epothilone ZK-219477, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well epothilone ZK-219477 works in treating patients with recurrent glioblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the therapeutic activity of epothilone ZK-219477 in patients with recurrent glioblastoma.

Secondary

* Determine the safety profile, mechanism of action, and pharmacokinetics of this drug in these patients.
* Gather information about the biological characteristics of the patients' tumor that may provide information on response or resistance to this drug.

OUTLINE: This is a nonrandomized, open-label, multicenter study.

Patients receive epothilone ZK-219477 IV over 3 hours on day 1. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

Blood samples are collected at baseline for biomarker analysis and for comparison of genetic alterations in tumor tissue with germline DNA. Blood samples are also collected periodically during course 1 for pharmacokinetic studies. Tumor tissue obtained at diagnosis, and possibly recurrence, is used for immunohistochemical analyses for biomarkers. Fluorescent in situ hybridization (FISH) is used to detect genetic alterations and gene expression.

After completion of study treatment, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed glioblastoma

  * Presence of oligodendroglial elements allowed provided they make up < 25% of tumor
* Measurable disease, defined as ≥ 1 bidimensionally measurable target lesion with a largest diameter of ≥ 2 cm by MRI within the past 2 weeks
* Recurrent disease

  * Documented by MRI after failing prior therapy (usually standard radiotherapy with concurrent and maintenance temozolomide)
  * Subsequent histologic confirmation of recurrence required for patients who received prior high-dose radiotherapy (> 65 Gy), stereotactic radiosurgery, or internal radiotherapy
* Multifocal disease that is not amenable to radiotherapy allowed provided the patient received no more than 1 line of prior chemotherapy

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin < 1.5 times upper limit of normal (ULN)
* AST and ALT < 2.5 times ULN
* Alkaline phosphatase < 2.5 times ULN
* Creatinine < 1.5 times ULN
* Clinically normal cardiac function
* No ischemic heart disease within the past 12 months

  * Stable ischemic heart disease (e.g., treated angina that is stable under appropriate therapy) allowed
* No New York Heart Association class III or IV cardiac insufficiency
* No unstable angina
* No arrhythmia
* No psychological, familial, sociological, or geographical factors that would preclude study compliance
* No other malignancy except cone-biopsied carcinoma of the cervix or adequately treated basal cell or squamous cell skin cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile female patients must use effective contraception during and for 3 months after completion of study treatment
* Fertile male patients must use effective contraception during and for 6 months after completion of study treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* More than 3 months since prior radiotherapy to the brain
* More than 3 months since prior surgery for recurrent primary brain tumor unless 1 of the following criteria are met:

  * Measurable residual disease documented by immediate (within 72 hours) postoperative imaging
  * Evidence of a progressive and measurable target lesion found at postoperative follow-up
  * Presence of a second measurable target lesion outside the surgical area
* Prior adjuvant temozolomide as first-line therapy allowed
* No prior chemotherapy for recurrent glioblastoma

  * One prior chemotherapy regimen given as adjuvant therapy allowed
* Concurrent corticosteroids allowed provided dose is stable or decreasing for ≥ 1 week
* No concurrent phenytoin, carbamazepine, or phenobarbital
* No concurrent Hypericum perforatum (St. John's wort)
* No concurrent enzyme-inducing antiepileptic drugs (EIAEDs)

  * Patients on EIAEDs should have been switched to non-EIAEDs with a wash-out period of ≥ 1 month
* No other concurrent anticancer agents (except alternative or homeopathic medicine)
* No other concurrent investigational treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-12; Primary Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Treatment success (complete or partial response or a progression-free survival at 6 months)

SECONDARY OUTCOMES:
Objective response
Duration of response
Toxicity
Progression-free survival at 6 months
Overall survival at 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Roger Stupp, MD, Study Chair — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

REFERENCES:
- [Result] Stupp R, Tosoni A, Bromberg JEC, Hau P, Campone M, Gijtenbeek J, Frenay M, Breimer L, Wiesinger H, Allgeier A, van den Bent MJ, Bogdahn U, van der Graaf W, Yun HJ, Gorlia T, Lacombe D, Brandes AA. Sagopilone (ZK-EPO, ZK 219477) for recurrent glioblastoma. A phase II multicenter trial by the European Organisation for Research and Treatment of Cancer (EORTC) Brain Tumor Group. Ann Oncol. 2011 Sep;22(9):2144-2149. doi: 10.1093/annonc/mdq729. Epub 2011 Feb 14. PMID 21321091
- [Result] Stupp R, Tosoni W, Taal W, et al.: Phase II trial of the epothilone analog sagopilone (ZK219477; ZK EPO) in patients with recurrent glioblastoma: initial report of the EORTC study 26061. [Abstract] J Clin Oncol 26 (Suppl 15): A-2015, 2008.